CLINICAL TRIAL: NCT05225389
Title: A Phase 1, Open-Label Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of a Single Oral Dose of [14C] CT1812 in Healthy Adult Male Subjects
Brief Title: Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of CT1812 in Healthy Adult Male Subjects
Acronym: COG0108
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: COG0108; SB1AG073028 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-02-04 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Carbon-14

STUDY DESIGN:
Intervention Model Description: Open-label, single-dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CT1812 (Experimental): Investigational Drug
  Interventions: Drug: 300 mg [C14] CT1812

INTERVENTIONS:
Drug: 300 mg [C14] CT1812 — Single dose of 300 mg CT1812 with microtracer dose of [C14]

SUMMARY:
Open-label, single-dose study to assess the absorption, metabolism, excretion and mass balance of [C14] CT1812

DETAILED DESCRIPTION:
Open-label, single-dose study to assess the absorption, metabolism, excretion and mass balance of [C14] CT1812 in 8 healthy male subjects

Subjects will be screened 28-days prior to dosing to determine eligibility.

Eligible subjects will be admitted to the clinical research unit (CRU) on Day -1. On Day 1, subjects will receive a single dose of CT1812 with a microtracer dose of [14C] CT1812. Whole blood, plasma, urine and fecal samples will be collection during the confinement period. Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

Subjects will be and discharged from the CRU following completion of procedures 168 hours post dose (Day 8)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male, 19 - 55 years of age
2. Male subjects must follow protocol specified contraception guidance as described in the protocol
3. Continuous non smoker who has not used tobacco/nicotine containing products for at least 3 months prior to dosing.
4. Body mass index (BMI) ≥18.0 and ≤30.0 kg/m2 at the Screening visit (subjects must not have experienced a weight loss or gain of >10% within 4 weeks of dosing).
5. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI/designee at the Screening visit.
6. History of a minimum of 1 bowel movement per day.
7. Able to swallow multiple capsules.
8. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Evidence of disease that, in the opinion of the PI/designee, may influence the outcome of the study within 4 weeks before dosing
2. Clinically significant illness, in the opinion of the PI/designee, that requires medical treatment within 8 weeks prior to dosing, or a clinically significant infection that requires medical treatment within 4 weeks prior to dosing.
3. Any history of GI surgery that may affect PK profiles of CT1812
4. Has evidence of a clinically significant abnormality in physical examination findings, vital signs, or clinical laboratory determinations at the Screening visit or Check-in.
5. Has a clinically significant ECG abnormality at the Screening visit or Check-in.
6. Estimated creatinine clearance <80 ml/min/1.73 m2 at the Screening visit.
7. Known history of clinically significant allergy to CT1812 or excipients at the Screening visit.
8. Has been diagnosed with acquired immune deficiency syndrome, or tests positive for human immunodeficiency virus (HIV), Hepatitis B virus surface antigen (HBsAg), or Hepatitis C virus (HCV) at the Screening visit.
9. Has a history of alcohol use disorder within the 2 years before the Screening visit.
10. Positive urine drug or alcohol results at the Screening visit or Check in.
11. Positive cotinine result at the Screening visit.
12. Unable to refrain from or anticipates the use of:

    * Any drugs, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to dosing except for those allowed in the protocol
    * Any drugs known to be significant inducers of CYP2D6 and CYP3A4 for 28 days prior to dosing.
13. Donation of blood or significant blood loss within 56 days prior to dosing.
14. Plasma donation within 7 days prior to dosing.
15. Poor peripheral venous access.
16. Recent history (within 2 weeks of Day 1) of abnormal bowel movements, such as diarrhea, loose stools, or constipation.
17. Has exposure to significant diagnostic or therapeutic radiation (e.g., serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in.
18. Has participated in a radiolabeled drug study where exposures are known to the PI within the previous 3 months prior to admission to the clinic for this study or participated in a radiolabeled drug study where exposures are not known to the PI within the previous 6 months prior to admission to the clinic for this study.
19. Has previously participated in a CT1812 investigational study.
20. Evidence or history of active suicidal thoughts in the 6 months preceding the screening visit; or have a history of a suicide attempt in the previous 2 years, or more than 1 lifetime suicide attempt; or are at serious suicide risk per the PIs clinical judgment.
21. Has any condition that would, in the opinion of the PI/designee or Sponsor, make the subject unsuitable for the study or is, in the opinion of the PI/designee, not likely to complete the study for any reason.
22. Participation in another clinical study within 30 days prior to dosing.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy, adult, males eligible for the study
Enrollment: 8 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Caggiano, MD, Study Director — Cognition Therapeutics Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were admitted to the clinical research unit (CRU).
Pre-assignment Details: Subjects were required to have a negative COVID-19 polymerase chain reaction (PCR) test in order to be enrolled in the study, as per the requirements outlined in the COVID-19 Clinical Pharmacology Unit Management Strategy and Study Risk Assessment documents.
Groups:
- 300 mg: Single oral dose of 300 mg CT1812 (2 capsules) with a microtracer dose of ~1 µCi [14C]-CT1812 (1 capsule).
Period: Overall Study
Arm/Group | 300 mg
Started | 8
Completed | 5
Not Completed | 3
Not completed — Three participants were discontinued by the Investigator on day 7 due to positive COVID-19 tests. | 3

BASELINE CHARACTERISTICS:
Arm/Group | 300 mg
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4
  White | 4
Weight [Mean (Standard Deviation); unit: Kg] | 81.91 (12.908)
Height [Mean (Standard Deviation); unit: cm] | 180.3 (3.54)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.233 (3.5198)

OUTCOME MEASURES:

1. Primary Outcome: Plasma CT1812 Concentration at 96 Hours Timepoint
Description: Plasma concentrations of CT1812 were determined using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) following a single oral dose of 300 mg (~1 μCi) [14C]-CT1812 administered in healthy adult male subjects.
Time Frame: Predose through 96 hours postdose
Population: For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of 0.00005 μg/mL are treated as 0.00 before the first quantifiable concentration and as missing elsewhere. No values were reported for the 120, 144, 168 hours timepoints. Three subjects were discontinued from the study after testing positive for COVID-19.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 300 mg
Number analyzed (Participants) | 8
μg/mL | 0.0000707 (0.0000240)

2. Primary Outcome: Plasma M6/CP199 Concentration at 144 Hours Timepoint
Description: Plasma concentrations of M6/CP199 were determined using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) following a single oral dose of 300 mg (~1 μCi) [14C]-CT1812 administered in healthy adult male subjects.
Time Frame: Predose through 144 hours postdose
Population: For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of 0.00005 μg/mL are treated as 0.00 before the first quantifiable concentration and as missing elsewhere. Three subjects were discontinued from the study after testing positive for COVID-19
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 300 mg
Number analyzed (Participants) | 8
μg/mL | 0.00001501 (0.0001370)

3. Primary Outcome: Plasma Total Radioactivity (TRA) Concentration CT1812-Equivalents at 168 Hours Timepoint
Description: Plasma Total Radioactivity Concentration of CT1812-Equivalents was performed using Liquid Scintillation Counting (LSC) method following a single oral dose of 300 mg (~1 μCi) [14C]-CT1812 administered in healthy adult male subjects.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours postdose
Population: For the calculation of summary statistics, values that are below the limits of quantitation (BLQ) ranging between 0.0261 - 0.0328 μg Eq/mL are treated as 0.00 before the first quantifiable concentration and as missing elsewhere. Three subjects were discontinued from the study after testing positive for COVID-19
Measure: Mean (Standard Deviation); unit: μg Eq/mL
Arm/Group | 300 mg
Number analyzed (Participants) | 8
μg Eq/mL | 0.08720 (0.068380)

4. Primary Outcome: Whole Blood Total Radioactivity (TRA) Concentration CT1812-Equivalents at 144 Hours Timepoint
Description: The analysis of Whole Blood Total Radioactivity Concentration of CT1812-Equivalents was performed using combustion followed by Liquid Scintillation Counting (LSC) method following a single oral dose of 300 mg (~1 μCi) [14C]-CT1812 administered in healthy adult male subjects.
Time Frame: Predose through 144 hours postdose
Population: For the calculation of summary statistics, values that are below the limits of quantitation (BLQ) ranging between 0.0368 - 0.0406 μg Eq/mL are treated as 0.00 before the first quantifiable concentration and as missing elsewhere. Three subjects were discontinued from the study after testing positive for COVID-19. No values were reported at 168 hours timepoint.
Measure: Mean (Standard Deviation); unit: μg Eq/mL
Arm/Group | 300 mg
Number analyzed (Participants) | 8
μg Eq/mL | 0.04413 (0.0086904)

5. Primary Outcome: Cumulative Percentage of Radioactive Dose (Cum%Dose) Excreted in the Urine
Description: Cumulative radioactive dose (Cum%Dose) excreted in the urine was determined using Liquid Scintillation Counting (LSC) following a single oral dose of 300 mg (~1 μCi) [14C]-CT1812 administered in healthy adult male subjects.
Time Frame: Predose and 0 to 4, 4 to 8, 8 to 12, and 12 to 24 hours postdose, and every 24 hours (pooled) until Day 8 (168 hours postdose).
Population: For the calculation of recovery parameters and summary statistics, concentration values that are below the limits.of quantitation (BLQ) ranging between 0.00205 to 0.00488 μg Eq/g are treated as 0.00. Three subjects were discontinued from the study after testing positive for COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of radioactive eliminated
Arm/Group | 300 mg
Number analyzed (Participants) | 8
percentage of radioactive eliminated | 81.13 (2.9789)

6. Primary Outcome: Cumulative Percentage of Radioactive Dose (Cum%Dose) Excreted in the Feces
Description: Cumulative radioactive dose (Cum%Dose) excreted in the feces was performed using combustion followed by Liquid Scintillation Counting (LSC) method following a single oral dose of 300 mg (~1 μCi) [14C]-CT1812 administered in healthy adult male subjects.
Time Frame: Predose, 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168 hours postdose
Population: For the calculation of recovery parameters and summary statistics of concentration data, concentration values that are below the limits of quantitation (BLQ) are treated as 0.00. Three subjects were discontinued from the study after testing positive for COVID-19.
Measure: Mean (Standard Deviation); unit: percentage of radioactive eliminated
Arm/Group | 300 mg
Number analyzed (Participants) | 8
percentage of radioactive eliminated | 19.29 (3,2123)

7. Primary Outcome: CT1812 Plasma Exposure According to AUC0-last Pharmacokinetic Parameter
Description: Plasma CT1812 Concentration were measured using the area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method following a single oral dose of 300 mg (~1 μCi) [14C]-CT1812 administered in healthy adult male subjects. Plasma concentrations of CT1812 were determined using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS).
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours postdose
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | 300 mg
Number analyzed (Participants) | 8
ug*hr/mL | 0.6636 (0.31014)

8. Primary Outcome: M6/CP199 Plasma Exposure According to AUC0-last Pharmacokinetic Parameter
Description: M6/CP199 Plasma Concentration was measured using the area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method following a single oral dose of 300 mg (~1 μCi) [14C]-CT1812 administered in healthy adult male subjects. M6/CP199 plasma concentrations were determined using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS).
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours postdose
Measure: Mean (Standard Deviation); unit: ug*hr/mL)
Arm/Group | 300 mg
Number analyzed (Participants) | 8
ug*hr/mL) | 48.46 (9.8619)

9. Primary Outcome: Plasma Total Radioactivity According to AUC0-last Pharmacokinetic Parameter
Description: Plasma Total Radioactivity was measured using the area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method following a single oral dose of 300 mg (~1 μCi) [14C]-CT1812 administered in healthy adult male subjects. Plasma Total Radioactivity Concentration of CT1812-Equivalents was performed using Liquid Scintillation Counting (LSC).
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours postdose
Measure: Mean (Standard Deviation); unit: μg Eq*hr/mL
Arm/Group | 300 mg
Number analyzed (Participants) | 8
μg Eq*hr/mL | 85.24 (11.436)

10. Primary Outcome: Whole Blood Total Radioactivity According to AUC0-last Pharmacokinetic Parameter
Description: Whole Blood Total Radioactivity was measured using the area under the concentration-time curve, from time 0 to the last observed non-zero concentration, as calculated by the linear trapezoidal method following a single oral dose of 300 mg (~1 μCi) [14C]-CT1812 administered in healthy adult male subjects. Plasma Total Radioactivity Concentration of CT1812-Equivalents was performed using Liquid Scintillation Counting (LSC)
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours postdose
Measure: Mean (Standard Deviation); unit: μg Eq*hr/mL
Arm/Group | 300 mg
Number analyzed (Participants) | 8
μg Eq*hr/mL | 52.51 (11.371)

11. Secondary Outcome: Whole Blood:Plasma Total Radioactivity Partitioning Ratios Over Time up to 144 Hours Timepoint
Description: This measure describes the percentage of TRA in whole blood relative to plasma. The fraction of [14C]-radioactivity associated with whole blood and plasma and with red blood cells and other cellular components of whole blood was determined by using the concentration of [14C]-radioactivity in whole blood and plasma.
Time Frame: Predose through 144 hours postdose
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 300 mg
Number analyzed (Participants) | 8
ratio | 0.4519 (0.11051)

12. Secondary Outcome: Number of TEAEs, Related TEAEs, SAEs, and Related SAEs
Description: Incidence and Severity of Adverse Events. All AEs that occurred during this clinical trial were coded using the Medical Dictionary for Regulatory Activities (MedDRA®), Version 24.1.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours
Population: Single oral dose of 300 mg CT1812 (2 capsules) with a microtracer dose of ~1 µCi [14C]-CT1812 (1 capsule).
Measure: Number; unit: Events
Arm/Group | 300 mg
Number analyzed (Participants) | 8
Events
  All TEAEs | 5
  Mild TEAEs | 3
  Moderate TEAEs | 2
  Severe TEAEs | 0
  Related TEAEs | 0
  TEAEs Leading to Treatment Discontinuation | 2

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | 300 mg
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg (N=8)
COVID 19 (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution will not publish or present any Study Data, results, Study Inventions, or Sponsor Confidential Information without prior written approval from the Sponsor. Institution will keep confidential and not disclose any information provided by or on behalf of Sponsor or CRO or that is generated, discovered, or obtained by any Party as a result of the Study (other than patient medical records), including the Study results, Study Inventions and information related thereto.

DOCUMENTS (2):
  • Study Protocol (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT05225389/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT05225389/SAP_001.pdf